CLINICAL TRIAL: NCT02218047
Title: An Open-label, Multicenter, Phase IIIb Study Assessing the Long-term Efficacy and Safety of AOP2014 and Standard First Line Treatment (BAT) in Patients With Polycythemia Vera Who Previously Participated in the PROUD-PV Study
Brief Title: AOP2014 vs. BAT in Patients With Polycythemia Vera Who Previously Participated in the PROUD-PV Study.
Acronym: CONTI-PV
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AOP Orphan Pharmaceuticals AG (Industry)
Collaborators: PharmaEssentia Corporation (for the U.S.) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CONTINUATION-PV; 2014-001357-17 (EudraCT Number)
Record Dates: First submitted 2014-08-14; First posted 2014-08-15 (Estimated); Last update posted 2021-06-01 (Actual); Status verified 2021-05

CONDITIONS: Polycythemia Vera
Keywords: Pegylated-Proline-interferon alpha-2b (AOP2014); Polycythemia Vera; PROUD-PV; CONTINUATION-PV; AOP Orphan; Polycythemia; Hematologic Diseases; Myeloproliferative Disorders; Bone Marrow Diseases; Interferon-alpha; Peginterferon alfa-2b
MeSH Terms: conditions — Polycythemia Vera; Polycythemia; Hematologic Diseases; Myeloproliferative Disorders; Bone Marrow Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Best available therapy (BAT) (Active Comparator): Best available therapy, as chosen by the investigator for patients who had been on HU in the 1 Year PROUD-PV study
  Interventions: Drug: Best available therapy (BAT)
- Pegylated-Proline-interferon alpha-2b (Experimental): AOP2014 for those patients who had been on AOP2014 in the PROUD-PV study
  Interventions: Drug: Pegylated-Proline-interferon alpha-2b

INTERVENTIONS:
Drug: Pegylated-Proline-interferon alpha-2b — Subjects will continue to receive the dosage which delivers the optimal disease response (hematocrit [Hct]<45%, platelets [PLTs]<400 x 109/L and leukocytes [WBCs]<10 x 109/L), as determined in the PROUD-PV study, preferably at the level of target blood values.
  Other Names: AOP2014
  Arms: Pegylated-Proline-interferon alpha-2b
Drug: Best available therapy (BAT) — Best available therapy as selected by the investigator
  Other Names: best available therapy
  Arms: Best available therapy (BAT)

SUMMARY:
Polycythemia Vera (PV) is a disease of bone marrow stem cells that manifests in a drastic increase of red blood cells and frequently also of white blood cells. The "thickening" of the blood in relation with a modified function of the cells has several consequences like increased blood pressure, pruritus of the skin, fatigue, disturbed blood circulation in the brain as well as fingers and toes and an increased risk of arterial and venous thrombosis (thrombosis is the formation of a blood clot in a vessel); like stroke, cardiac infarction, deep vein thrombosis in the legs. In case of a strong increase of platelets there is an additional risk of bleedings. As the disease progresses the size of spleen and liver increased in most cases and the bone marrow shows signs of fibrosis. In some cases of PV a progression at a later time point to a leukemia (increased formation of white blood cells) can occur.

The aim of this study is to show that the study drug AOP2014 (pegylated proline interferon alpha-2b) has the long term efficacy and safety in controlling the disease. A comparison arm is receiving best available therapy as selected by the investigator. Response to the treatment is measured by several blood parameters as well as size of the spleen.

Interferon-alpha has been shown to be effective in controlling the blood parameters by immunologically influencing the blood building cells. This can lead to a suppression of the disease-causing stem cells and help healthy stem cells to proliferate. Through this mechanism it is possible that Interferon-alpha can avoid long-term damaging effects of the disease.

DETAILED DESCRIPTION:
This is a Phase III, parallel-arm, open-label continuation of the PROUD-PV study performed in adults diagnosed with Polycythemia Vera (PV). Patients who received AOP2014 in the primary study, PROUD-PV will continue on AOP2014, patients who received HU in the PROUD-PV study will receive best available therapy as selected by the investigator. Only patients who completed PROUD-PV including the end of study visit will be enrolled into this continuation study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who completed the 12 months AOP2014 treatment arm of the PROUD-PV study and at the "end-of-treatment visit" (EoT) of the PROUD-PV study who fulfill at least one of the following criteria:

   * normalization of at least two out of three main blood parameters (Hct, PLTs and WBCs) if these parameters were moderately increased (Hct<50%, WBC<20 x 109/L, PLTs<600 x 109/L) at baseline of the PROUD-PV study, OR
   * >35% decrease of at least two out of three main blood parameters (Hct, PLTs and WBCs) if these parameters were massively increased (Hct>50%, WBCs>20 x 109/L, PLTs>600 x 109/L), at baseline of the PROUD-PV study, OR
   * normalization of spleen size, if spleen was enlarged at baseline of the PROUD-PV study, OR
   * otherwise a clear, medically verified benefit from treatment with AOP2014 (e.g. normalization of disease-related micro-vasculatory symptoms, substantial decrease of JAK2 allelic burden).
2. Signed written ICF.

Exclusion criteria:

Withdrawal criteria, as specified in the PROUD-PV study, which mandate treatment discontinuation:

1. Non-recovery from the AOP2014 related toxicities to the grade (usually, Grade I) which allows continuation of the treatment.
2. HADS score of 11 or higher on either or both of the subscales, and /or development or worsening of the clinically significant depression or suicidal thoughts.
3. Progressive and clinically significant increase of liver enzyme levels despite dose reduction, or if such increase is accompanied by increased bilirubin level, any signs or symptoms of a clinically significant autoimmune disease.
4. Clinically significant development of a new ophthalmologic disorder, or worsening of a pre-existing one, during the study.
5. Loss of efficacy of AOP2014 or any comparable situation where no further benefits of treatment continuation are expected by the investigator.

The main efficacy evaluation criterion will be disease response defined as Hct<45% without phlebotomy (at least 3 months since the last phlebotomy), PLTs<400 x 109/L, WBCs<10 x 109/L, and normal spleen size.

The main efficacy endpoint will be the maintenance rate of disease response at assessment visits (every three months).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2021-04-29 (Actual); Study Completion 2021-04-29 (Actual)

PRIMARY OUTCOMES:
Disease response at quarterly assessment visits | 3 years
  The primary efficacy endpoint will be the rate of disease response at assessment visits (every 3 months).
  The co-primary efficacy evaluation criterion will be (1) disease response defined as hematologic response: Hct<45% without phlebotomy (at least 3 months since the last phlebotomy), PLTs<400 x 109/L, WBCs<10 x 109/L, and normal spleen size, and (2) disease response defined as hematologic response (Hct<45% without phlebotomy (at least 3 months since the last phlebotomy), PLTs<400 x 109/L, WBCs<10 x 109/L), resolution and/or clinically improvement of disease-related signs (clinical significant splenomegaly) and disease-related symptoms (microvascular disturbances, pruritus, headache).

CONTACTS AND LOCATIONS:
Overall Officials: Heinz Gisslinger, MD, Principal Investigator — Med Uni Wien
Locations (47):
- Austria (7):
  - LKH Graz, Graz
  - University Hospital Innsbruck, Innsbruck
  - Elisabethinen Hospital Linz, Linz
  - Salzburg Regional Hospital, Salzburg
  - Hanusch Hospital, Vienna
  - Medical University Vienna, Vienna
  - Hospital Wels-Grieskirchen, Wels
- Bulgaria (4):
  - University Multiprofile Hospital for Active Treatment "Sveti Georgi", Plovdiv, Plovdiv
  - Specialized Hospital for Active Treatment of Hematological Diseases, Sofia
  - Multiprofile Hospital for Active Treatment "Sveta Marina", Varna, Varna
  - Multiprofile Hospital for Active Treatment - Hristo Botev, Vratsa, First Department of Internal Medicine, Vratsa
- Czechia (4):
  - University Hospital Brno, Brno
  - University Hospital Hradec Kralove, Hradec Králové
  - University Hospital Kralovske Vinohrady, Prague
  - University Hospital Motol, Prague
- France (3):
  - Institute Paoli-Calmettes, Marseille
  - Hospital Saint-Louis, Paris
  - Clinical Research Center CIC, Poitiers
- Germany (3):
  - Aachen University Hospital, Medical Clinic IV, Aachen
  - University Hospital Bonn, Center for Internal Medicine, Medical Clinic and Outpatient Clinic III, Bonn
  - University Hospital Carl Gustav Carus, Medical Clinic and Polyclinic I, Dresden
- Hungary (5):
  - St Istvan and St Laszlo Hospital of Budapest, Budapest
  - University of Debrecen, Debrecen
  - Bekes County Pandy Kalman Hospital, 1st Department of Medicine, Hematology, Gyula
  - Kaposi Mor County Teaching Hospital, Kaposvár
  - University of Szeged, Albert Szent-Gyorgyi Clinical Center, Koranyi fasor 6, Szeged
- Poland (5):
  - University Hospital in Cracow, Krakow
  - Independent Public Teaching Hospital No.1 in Lublin, Lublin
  - Fryderyk Chopin Provincial Specialized Hospital, Rzeszów
  - Nicolaus Copernicus Municipal Specialist Hospital, Torun
  - Institute of Hematology and Transfusion Medicine, Warsaw
- Romania (3):
  - Emergency Clinical County Hospital Brasov, Brasov
  - Bucharest University Emergency Hospital, Bucharest
  - Coltea Clinical Hospital, Bucharest
- Russia (5):
  - Baranov Republican Hospital, Petrozavodsk
  - Samara Kalinin Regional Clinical Hospital, Samara
  - Komi Republican Oncology Center, Syktyvkar
  - Tula Regional Clinical Hospital, Tula
  - Yaroslavl Regional Clinical Hospital, Yaroslavl
- Slovakia (2):
  - University Hospital with Outpatient Clinic F.D. Roosevelt, Banská Bystrica
  - Saint Cyril and Metod University Hospital Bratislava, Bratislava
- Hospital del Mar, Barcelona, Spain
- Ukraine (5):
  - Cherkasy Regional Oncology Center, Regional Treatment and Diagnostics Hematology Center, Cherkasy
  - Dnipropetrovsk City Multispecialty Clinical Hospital #4, Dnipropetrovsk
  - National Research Center for Radiation Medicine, Institute of Clinical Radiology, Kiev
  - Institute of Blood Pathology and Transfusion Medicine, Lviv
  - O.F. Herbachevskyi Regional Clinical Hospital, Zhytomyr